CLINICAL TRIAL: NCT03800381
Title: Pharmacokinetics of Anti-tuberculosis and Antiretroviral Drugs in Children
Brief Title: Adequacy of the New Pediatric Isoniazid/Rifampin/Pyrazinamide (HRZ) Tablet
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB201801820 - HRZ PK -N; 5R01HD071779-11 (NIH)
Record Dates: First submitted 2019-01-03; First posted 2019-01-11 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Tuberculosis; Human Immunodeficiency Virus; Coinfection
Keywords: Pharmacokinetic; Pharmacogenomic; Antituberculosis drugs; Children; Tuberculosis; TB/HIV coinfection
MeSH Terms: conditions — Tuberculosis; Acquired Immunodeficiency Syndrome; Coinfection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Ethylenediaminetetraacetic acid (EDTA) plasma and whole blood deoxyribonucleic acid (DNA)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Active TB only: Children with clinical diagnosis or acid-fast bacilli (AFB) smear positive TB disease
  Interventions: Other: Observational PK study
- Active TB with HIV Co-infection: Children with clinical diagnosis or AFB smear positive TB disease who test positive for HIV infection
  Interventions: Other: Observational PK study

INTERVENTIONS:
Other: Observational PK study — The study team will examine the PK and tolerability of the new HRZ 50/75/150 mg dispersible tablet in children with TB with and without HIV coinfection. Intensive PK testing will be performed after at least 4 weeks of treatment in children on first-line anti-TB therapy using the new pediatric HRZ FDC tablet.
  Other Names: New pediatric isoniazid/rifampin/pyrazinamide (HRZ) FDC tablet

SUMMARY:
Lack of quality-assured pediatric formulations of the first-line antituberculosis (anti-TB) drugs is barrier to optimized tuberculosis (TB) treatment outcome in children. In 2010 and subsequently modified in 2014, the World Health Organization (WHO) recommended increased dosages of the first-line anti-TB drugs for children, but there were no child-friendly fixed-dose combination (FDC) formulations based on the guidelines. A large proportion of children treated with the new guidelines using old formulations did not achieve the desired rifampin peak concentration (Cmax) > 8 mg/L and pyrazinamide Cmax > 35 mg/L. The TB Alliance and the WHO led the development of a new child-appropriate isoniazid/rifampin/pyrazinamide (HRZ) and isoniazid/rifampin (HR) FDC formulation in line with current WHO recommended dosing guidelines. The new formulations dissolve quickly in liquid, have palatable fruit flavors, and are expected to improved daily adherence but no studies have evaluated the pharmacokinetics (PK) of the FDC formulation in children. The study team hypothesize that the new dispersible HRZ FDC tablet, dosed according to current WHO weight-band dosing recommendations will result in better PK parameters for each drug component than that achieved by the old formulation.

DETAILED DESCRIPTION:
This study will evaluate the PK of the new pediatric HRZ FDC tablet in Ghanaian children with TB with and without HIV coinfection. The new HRZ FDC dispersible tablet was designed to be child-friendly and to achieve recommended dosages for each weight-band. The formulation has been rolled out in Africa without PK studies in the target population to verify that the tablets achieves adequate drug concentrations. The current study will evaluate the adequacy of the formulation by examining the PK of the component drugs as well as the effect of HIV coinfection. The direct PK data will be used in a population PK model and stimulations to define optimal weight-band dosages and proportions of the components of the pediatric FDC tablets.

ELIGIBILITY:
Inclusion Criteria:

* Children with active TB with or without HIV coinfection. Active TB diagnosis defined by clinical criteria consistent with active TB and/or a positive AFB smear.
* Available for follow-up until completion of TB treatment and/or achievement of a study endpoint like discontinuation of therapy, and/or pharmacokinetic sampling.

Exclusion Criteria:

* Children with concurrent conditions other than HIV, have acute hepatitis within 30 days of study entry, persistent vomiting, and diarrhea will be excluded from the study.
* Unable to obtain informed signed consent from parent(s) or legal guardian.
* Have AIDS-related opportunistic infections other than TB, history of or proven acute hepatitis within 30 days of study entry, persistent vomiting, or diarrhea.
* Hemoglobin < 6 g/dl, white blood cells < 2500/mm3, serum creatinine > 1.5 mg/dl, aspartate transaminase (AST) and alanine transaminase (ALT) > 2 times upper limit of normal.

Ages: 3 Months to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 3 months to14 years with active TB with or without HIV co-infection
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Peak concentration (Cmax) of isoniazid, rifampin and pyrazinamide in the new pediatric HRZ FDC tablet. | After at least 4 weeks of anti-TB therapy
  Mean and median Cmax of rifampin, isoniazid and pyrazinamide in children with TB treated with the new HRZ FDC tablet.
Area under the time-concentration curve from 0-8 hours (AUC0-8h) of isoniazid, rifampin and pyrazinamide in the new pediatric HRZ FDC tablet. | After at least 4 weeks of anti-TB therapy
  Mean and median AUC0-8h of rifampin, isoniazid and pyrazinamide in children with TB treated with the new HRZ FDC tablet.
Cmax of isoniazid, rifampin and pyrazinamide in children with TB with and without HIV coinfection | After at least 4 weeks of anti-TB therapy
  Geometric mean values of Cmax of rifampin, isoniazid and pyrazinamide in children with HIV/TB coinfection compared to those with TB alone.
AUC0-8h of isoniazid, rifampin and pyrazinamide in children with TB with and without HIV coinfection. | After at least 4 weeks of anti-TB therapy
  Geometric mean values of AUC0-8h of rifampin, isoniazid and pyrazinamide in children with HIV/TB coinfection compared to those with TB alone.

SECONDARY OUTCOMES:
AUC0-8h of isoniazid, rifampin and pyrazinamide in the new versus old pediatric HRZ FDC tablet. | After at least 4 weeks of anti-TB therapy
  Geometric mean values of AUC0-8h of rifampin, isoniazid, and pyrazinamide in children with TB treated with the new FDC tablet compared to those treated with the old formulation in our previous study (historical controls).
Cmax of isoniazid, rifampin and pyrazinamide in the new versus old pediatric HRZ FDC tablet. | After at least 4 weeks of anti-TB therapy
  Geometric mean values of Cmax of rifampin, isoniazid, and pyrazinamide in children with TB treated with the new FDC tablet compared to those treated with the old formulation in our previous study (historical controls).
Proportion of children treated with new pediatric HRZ FDC tablet who develop with liver enzymes elevations. | After at least 4 weeks of anti-TB therapy
  Frequency of liver enzymes elevations compared to baseline requiring treatment modification in children with TB with and without HIV coinfection.
Identify optimal weight-band dosages of the new HRZ FDC tablet | After at least 4 weeks of anti-TB therapy
  Use a population PK model that incorporates demographic, clinical and genetic factors and stimulations to identify the optimal weight-band dosing of the new FDC formulation.

CONTACTS AND LOCATIONS:
Overall Officials: Awewura Kwara, MD, Principal Investigator — University of Florida
Locations (1):
- Kwame Nkrumah University of Science and Technology, Kumasi, Ghana

IPD SHARING:
Plan to Share IPD: Undecided